CLINICAL TRIAL: NCT00053053
Title: A Double-Blind Study Of Nutritional Intervention For The Treatment Of Cancer Cachexia Using Juven® Nutritional Supplement
Brief Title: Comparison of Nutritional Supplements in Preventing Weight Loss in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RTOG-0122; CDR0000269100
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2013-10

CONDITIONS: Cachexia; Lymphoma; Lymphoproliferative Disorder; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; cachexia; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; intraocular lymphoma; AIDS-related peripheral/systemic lymphoma; recurrent adult Burkitt lymphoma; anaplastic large cell lymphoma; post-transplant lymphoproliferative disorder; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Cachexia; Lymphoma; Lymphoproliferative Disorders; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Intraocular Lymphoma; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Juven supplement (Experimental): Juven nutritional supplement given twice a day for 8 weeks
  Interventions: Dietary Supplement: Juven
- Non-Juven supplement (Active Comparator): Non-Juven nutritional supplement given twice a day for 8 weeks
  Interventions: Dietary Supplement: Non-Juven Supplement

INTERVENTIONS:
Dietary Supplement: Juven
  Arms: Juven supplement
Dietary Supplement: Non-Juven Supplement
  Arms: Non-Juven supplement

SUMMARY:
RATIONALE: Nutritional supplements may help prevent loss of appetite, weight loss, and fatigue in patients with advanced cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two nutritional supplements in preventing loss of appetite, weight loss, and fatigue in patients who have stage III or stage IV solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the change in lean body mass of patients treated with Juven® vs a non-Juven® supplement.
* Compare the change in fatigue and quality of life of patients treated with these supplements.
* Compare the results of plethysmography, bioimpedance, and skinfold measurement in patients treated with these supplements.
* Compare the weight change in patients treated with these supplements.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to primary disease site (lung vs others), concurrent chemotherapy (yes vs no), evidence of metastases (yes vs no), and degree of weight loss (2-5% vs 6-10%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral Juven® supplement twice daily for 8 weeks.
* Arm II: Patients receive oral non-Juven® supplement twice daily for 8 weeks. All patients undergo lean body mass measurement (to include multiple body composition and weight change) and fatigue and quality of life assessments at baseline and then at 4 and 8 weeks.

PROJECTED ACCRUAL: A total of 468 patients (234 per treatment arm) will be accrued for this study within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor or lymphoma with no leukemic aspect

  * Stage III or IV or any other stage associated with current metastatic disease at presentation
  * No primary or metastatic brain tumors
* Weight loss of at least 2% but no more than 10% within the past 3 months
* No ascites

PATIENT CHARACTERISTICS:

Age

* 17 and over

Performance status

* Zubrod 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* No hypercalcemia

Cardiovascular

* No persistent moderate or severe peripheral edema
* No uncontrolled congestive heart failure

Gastrointestinal

* No enteric fistula
* No concurrent intestinal obstruction

  * Prior intestinal obstruction allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* No uncontrolled infections
* No other serious medical illness
* No metabolic disorder

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Concurrent chemotherapy allowed

Endocrine therapy

* No dexamethasone as an appetite stimulant
* Intermittent dexamethasone during concurrent chemotherapy allowed

Radiotherapy

* Concurrent radiotherapy allowed

Surgery

* At least 1 week since prior minor surgery
* At least 3 weeks since prior major surgery

Other

* At least 30 days since prior total parenteral nutrition
* No concurrent parenteral feedings
* No concurrent known appetite stimulants (e.g., megestrol or dronabinol)
* No concurrent omega 3 fatty acids or their congeners (e.g., ProSure™)
* No concurrent amino acid supplements
* Concurrent use of other dietary supplements (e.g., Ensure® or Boost) is allowed
* Concurrent enteral feedings via PEG or nasogastric tube are allowed

Ages: 17 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2002-12; Primary Completion 2005-03 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Lean body mass | Study entry to 8 weeks

SECONDARY OUTCOMES:
Fatigue | Study entry to 8 weeks
Quality of Life | Study entry to 8 weeks
Body weight | Study entry to 8 weeks
Correlation between change in lean body mass and body plethysmography, bioimpedance and skin-fold measurement | Study entry to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence B. Berk, MD, PhD, Study Chair — CCOP - Columbus
Locations (250):
- United States (230):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Comprehensive Cancer Institute, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Montgomery Cancer Center, Montgomery, Alabama
  - DCH Cancer Treatment Center, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Regional Cancer Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center at Huntington Hospital, Pasadena, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - Radiation Oncology Centers - Sacramento, Sacramento, California
  - Radiation Medical Group, Incorporated, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - St. Joseph's Regional Cancer Center, Stockton, California
  - Torrance Memorial Medical Center, Torrance, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - 21st Century Oncology - Fort Myers, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Florida Radiation Oncology Group, Jacksonville, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Cancer Center at St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Oncology Institute of Greater Lafayette, Lafayette, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Esther Marie Hatton Cancer Care Center at St. Elizabeth Medical Center, Edgewood, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Cancer Center at Lexington Clinic, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Louisville Radiation Oncology Center at Caritas Regional Cancer Center, Louisville, Kentucky
  - Merle M. Mahr Cancer Center at Regional Medical Center of Hopkins County, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center - Bramhall Campus, Portland, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Cancer Center at Greater Baltimore Medical Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - William Beaumont Hospital - Troy Campus, Troy, Michigan
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program - Marlton, Mount Holly, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center - Mainland Division, Pomona, New Jersey
  - University Medical Center at Princeton, Princeton, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - South Jersey Healthcare Regional Cancer Center, Vineland, New Jersey
  - Associated Radiologists, P.A. at Warren Radiation Therapy Center, Warren Township, New Jersey
  - Radiation Oncology Associates, PA, Albuquerque, New Mexico
  - Lourdes Regional Cancer Center, Binghamton, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Finger Lakes Radiation Oncology Center at Clifton Springs Hospital and clinic, Clifton Springs, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - North Shore Radiation Oncology, Setauket, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Akron City Hospital at Summa Health System, Akron, Ohio
  - Cancer Center at Christ Hospital, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Frank C. Love Cancer Institute at St. Anthony Hospital, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - LaFortune Cancer Center at St. John Health System, Tulsa, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - John and Dorothy Morgan Cancer Center at Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes-Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Cancer Center at Wellspan Health, York, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Arlington Cancer Center - Arlington, Arlington, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Bon Secours Cancer Care at St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Cancer Institute at Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia St. Mary's - Columbia Campus, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at St. Luke's Medical Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (20):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre at Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - CHUS-Hopital Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Berk L, James J, Schwartz A, Hug E, Mahadevan A, Samuels M, Kachnic L; RTOG. A randomized, double-blind, placebo-controlled trial of a beta-hydroxyl beta-methyl butyrate, glutamine, and arginine mixture for the treatment of cancer cachexia (RTOG 0122). Support Care Cancer. 2008 Oct;16(10):1179-88. doi: 10.1007/s00520-008-0403-7. Epub 2008 Feb 22. PMID 18293016